CLINICAL TRIAL: NCT04459286
Title: A Randomized, Open Label Trial to Investigate the Efficacy and Safety of Nitazoxanide Plus Atazanavir/Ritonavir for the Treatment of COVID-19: a Pilot Study
Brief Title: The Nitazoxanide Plus Atazanavir for COVID-19 Study
Acronym: NACOVID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IDSMB recommendation
Sponsor: Obafemi Awolowo University (Other)
Collaborators: University of Liverpool (Other); African Centre of Excellence for Genomics of Infectious Diseases (Unknown); Infectious Disease Hospital Olodo (Unknown); Obafemi Awolowo University Teaching Hospitals Complex (Unknown); Osun State Ministry of Health (Unknown); Olabisi Onabanjo University Teaching Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NACOVID
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Covid-19
Keywords: SARS-CoV infection; COVID-19; coronavirus
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — nitazoxanide; Atazanavir Sulfate; Ritonavir; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Participants in this arm will receive SOC alone, which will be as determined by the clinical team at the treatment centres in line with the current National Interim Guidelines for Clinical Management of COVID-19
  Interventions: Other: Standard of Care
- SOC plus Intervention (Experimental): Participants in this arm will receive SOC plus study intervention composed of orally administered nitazoxanide and atazanavir/ritonavir tablets
  Interventions: Drug: Nitazoxanide and atazanavir/ritonavir; Other: Standard of Care

INTERVENTIONS:
Drug: Nitazoxanide and atazanavir/ritonavir — 1000 mg nitazoxanide tablets twice daily and 300/100 mg atazanavir/ritonavir tablets once daily with meal
  Arms: SOC plus Intervention
Other: Standard of Care — SOC will be as determined by the clinical team at the treatment centres in line with the current National Interim Guidelines for Clinical Management of COVID-19

SUMMARY:
Since the outbreak of the novel coronavirus disease in 2019 (COVID-19), an unprecedented global search for potential therapeutics and vaccines is ongoing. In this study, a combination of two drugs that have been shown to be effective against the germ that causes COVID-19 in the laboratory will be tested in patients diagnosed with moderate to severe COVID-19. One of the drugs is called nitazoxanide and the second is atazanavir/ritonavir. Nitazoxanide has been used for the treatment of diarrhea since 2004 while atazanavir/ritonavir was approved for HIV treatment in 2003. They are known to be safe in humans.

In this pilot study, 98 COVID-19 patients will be recruited into two groups. The 49 patients in group 1 will receive the standard of care determined by their primary care providers while the 49 patients in group 2 will receive both the standard of care combined with the two study drugs. Patients in group 2 will receive the study drugs for 14 days and all patients will be monitored for a total of 28 days.

The time it takes for the germ that causes COVID-19 to be completely removed from the body (in nasal secretions) and the time to clinical improvement will be monitored in all patients and compared between the two groups.

DETAILED DESCRIPTION:
COVID-19 caused by a novel severe acute respiratory syndrome coronavirus (SARS-CoV-2) is an unprecedented global public health challenge which as at July 1, 2020 has spread to over 210 countries with over 10.6 million cases resulting in 514,808 deaths. More than 1500 clinical trials are currently ongoing in an unprecedented global search for potential therapeutics and vaccines. With increasing number of cases reported in low- and middle-income countries and and the possibility of a second wave of infections in countries where the pandemic appears to have slowed, studies to investigate promising therapies are urgently needed, especially those that can significantly reduce time to viral clearance and mortality. Shortening SARS-CoV-2 clearance time will lower treatment cost and reduce the economic impact of the pandemic.

The purpose of this phase 2 trial is to investigate the efficacy and safety of repurposed antiprotozoal and antiretroviral drugs, nitazoxanide and atazanavir/ritonavir, in achievement of SARS-CoV-2 PCR negativity and shorten the time to clinical improvement in patients diagnosed with moderate to severe COVID-19. The selection of candidates for this COVID-19 drug repurposing trial was guided by three pharmacological considerations: (1) demonstration of in-vitro anti-SARS-CoV-2 activity at doses shown or predicted to be tolerated by humans, (2) the feasibility of achieving effective concentration in relevant compartments, and (3) established human safety record.

This is a pilot phase 2, open label randomized controlled trial. A total of 98 patients with confirmed COVID-19 diagnosis (defined as SARS-CoV-2 polymerase chain reaction (PCR) positive nasopharyngeal swab) will be recruited from participating treatment centres. Participants will be randomised to receive either the standard of care (SOC) plus nitazoxanide for 14 days, starting from day 1 or the SOC alone for 14 days.

Participants will be recruited within 2 days of admission into COVID-19 treatment centre. Before enrollment, they will be given adequate information about the trial, opportunity to ask questions, and sufficient time to consider participation. Before any screening procedures, a written consent will be obtained from each eligible subject who agrees to participate in the trial. Participants will then be randomly allocated 1:1 to receive either the SOC alone (control group) or SOC plus study drug (intervention group). Parallel assignment will be used to prevent sample size imbalance between groups and control for important covariates (e.g. age, comorbidities, gender) that may affect trial results. Participants in the intervention group will receive 1000 mg nitazoxanide (two tablets of 500 mg each) with meal two times daily (8 am and 8 pm) and one tablet of 300/100 mg atazanavir/ritonavir with meal once daily (8 pm) in addition SOC. Participants in the control arm will receive the SOC alone. SOC will be as determined by the clinical team at the treatment centres in line with the current National Interim Guidelines for Clinical Management of COVID-19.

The treatment duration for participants in the intervention group will be 14 days. However, follow up will continue until day 28 after study entry at the end of which all participants will exit the study. Evaluations at follow up visits will include daily symptoms monitoring using inFLUenza Patient-Reported Outcome (FLU-PRO) questionnaire, daily vitals, daily clinical improvement assessment, and swab and/or sputum collection for SARS-CoV-2 on days 2, 4, 6, 7, 14, and 28.

Sample size estimation is based on the assumption that an improvement of at least 60-80% in time to SARS-CoV-2 PCR negativity and symptoms resolution can be achieved in the intervention group compared with the control group. Hence, a total sample size of 89 will provide at least 80% power to show or exclude 60% improvement in time to SARS-CoV-2 PCR negativity. This assumes a two-sided and 5% type 1 error rate. Therefore, providing for a 10% loss to follow up rate, a total of 98 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide written informed consent
* At least 18 and not more than 75 years of age at study entry
* SARS-CoV-2 infection confirmed by PCR test within 4 days before randomization
* Currently symptomatic (fever or chills, cough, myalgia, sore throat, shortness of breath, or new onset of anosmia or ageusia) and at COVID-19 isolation and treatment centre

Exclusion Criteria:

* Inability to take orally administered medication or food
* Known hypersensitivity to study medication
* Pregnant or lactating (unless practicing exclusive replacement feeding for the entire study duration)
* Participation in any other interventional trial for COVID-19 (observational study co-enrollment allowed)
* Concurrent treatment with other agents with actual or possible direct-acting antiviral activity against SARS-CoV-2 less than 24 hours prior to study drug dosing
* Concurrent use of agents with known or uncertain interaction with study drugs, including ritonavir
* Requiring mechanical ventilation at screening
* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) above 5 times upper limit of normal (ULN)
* Creatinine clearance below 50 mL/min using the Cockcroft-Gault formula for participants above 18 years of age

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-02 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | 28 days
  Proportion of patients with clinical improvement, as defined by live discharge from the hospital, a decrease of at least 2 points from baseline on a 7-point ordinal scale, or both.
Time to SARS-CoV-2 negativity | 28 days
  Proportion of participants with SARS-CoV-2 polymerase chain reaction (PCR) negative result at Days 7, 10, 14 and 28
Difference in SARS-CoV-2 AUC | 28 days
  Temporal patterns of SARS-CoV-2 viral load quantified by RT-PCR from nasal swabs or sputum of patients receiving SOC alone versus SOC plus study drug

SECONDARY OUTCOMES:
Time to symptoms resolution | 28 days
  Time to symptoms resolution as monitored by the Performance of the inFLUenza Patient-Reported Outcome (FLU-PRO) questionnaire with some modifications for COVID-19
Clinical status as assessed with the seven-category ordinal scale on days 7 and 14 | 14 days
Duration of hospitalization in survivors | 28 days
Day 28 mortality | 28 days
Time from treatment initiation to death | 28 days
Proportion with viral RNA detection over time | 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- Nigeria (2):
  - Olabisi Onabanjo University Teaching Hospital, Sagamu, Ogun State
  - Infectious Disease Hospital, Olodo, Ibadan, Oyo State

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossignol JF. Nitazoxanide, a new drug candidate for the treatment of Middle East respiratory syndrome coronavirus. J Infect Public Health. 2016 May-Jun;9(3):227-30. doi: 10.1016/j.jiph.2016.04.001. Epub 2016 Apr 16. PMID 27095301
- [Background] Cao J, Forrest JC, Zhang X. A screen of the NIH Clinical Collection small molecule library identifies potential anti-coronavirus drugs. Antiviral Res. 2015 Feb;114:1-10. doi: 10.1016/j.antiviral.2014.11.010. Epub 2014 Nov 28. PMID 25451075
- [Background] Haffizulla J, Hartman A, Hoppers M, Resnick H, Samudrala S, Ginocchio C, Bardin M, Rossignol JF; US Nitazoxanide Influenza Clinical Study Group. Effect of nitazoxanide in adults and adolescents with acute uncomplicated influenza: a double-blind, randomised, placebo-controlled, phase 2b/3 trial. Lancet Infect Dis. 2014 Jul;14(7):609-18. doi: 10.1016/S1473-3099(14)70717-0. Epub 2014 May 19. PMID 24852376
- [Background] Arshad U, Pertinez H, Box H, Tatham L, Rajoli RKR, Curley P, Neary M, Sharp J, Liptrott NJ, Valentijn A, David C, Rannard SP, O'Neill PM, Aljayyoussi G, Pennington SH, Ward SA, Hill A, Back DJ, Khoo SH, Bray PG, Biagini GA, Owen A. Prioritization of Anti-SARS-Cov-2 Drug Repurposing Opportunities Based on Plasma and Target Site Concentrations Derived from their Established Human Pharmacokinetics. Clin Pharmacol Ther. 2020 Oct;108(4):775-790. doi: 10.1002/cpt.1909. Epub 2020 Jun 14. PMID 32438446
- [Background] Rajoli RK, Pertinez H, Arshad U, Box H, Tatham L, Curley P, Neary M, Sharp J, Liptrott NJ, Valentijn A, David C, Rannard SP, Aljayyoussi G, Pennington SH, Hill A, Boffito M, Ward SA, Khoo SH, Bray PG, O'Neill PM, Hong WD, Biagini G, Owen A. Dose prediction for repurposing nitazoxanide in SARS-CoV-2 treatment or chemoprophylaxis. medRxiv [Preprint]. 2020 May 6:2020.05.01.20087130. doi: 10.1101/2020.05.01.20087130. PMID 32511548
- [Derived] Fowotade A, Bamidele F, Egbetola B, Fagbamigbe AF, Adeagbo BA, Adefuye BO, Olagunoye A, Ojo TO, Adebiyi AO, Olagunju OI, Ladipo OT, Akinloye A, Onayade A, Bolaji OO, Rannard S, Happi C, Owen A, Olagunju A. A randomized, open-label trial of combined nitazoxanide and atazanavir/ritonavir for mild to moderate COVID-19. Front Med (Lausanne). 2022 Sep 8;9:956123. doi: 10.3389/fmed.2022.956123. eCollection 2022. PMID 36160134
- [Derived] Olagunju A, Fowotade A, Olagunoye A, Ojo TO, Adefuye BO, Fagbamigbe AF, Adebiyi AO, Olagunju OI, Ladipo OT, Akinloye A, Adeagbo BA, Onayade A, Bolaji OO, Happi C, Rannard S, Owen A. Efficacy and safety of nitazoxanide plus atazanavir/ritonavir for the treatment of moderate to severe COVID-19 (NACOVID): A structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Jan 4;22(1):3. doi: 10.1186/s13063-020-04987-8. PMID 33397457
- See also: Nitaxoxanide Prescribing Information — https://www.accessdata.fda.gov/drugsatfda_docs/label/2016/021497s001,021498s004lbl.pdf
- See also: Atazanavir inhibits SARS-CoV-2 replication and pro-inflammatory cytokine production — https://www.biorxiv.org/content/10.1101/2020.04.04.020925v2
- See also: Atazanavir/ritonavir Prescribing Information — https://www.accessdata.fda.gov/drugsatfda_docs/label/2011/021567s026lbl.pdf